CLINICAL TRIAL: NCT06893055
Title: Strength-Endurance Circuit Training in Parkinson's Disease: Effects on Disease Severity, Physical Performance, Blood Biomarkers and Quality of Life.
Brief Title: Strength-Endurance Circuit Training in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Jakub Vítek, Physiotherapist, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 56125
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Parkinson Disease; Strength training; Endurance training; Physiotherapy; Irisin; Quality of Life; Physical performance
MeSH Terms: conditions — Parkinson Disease | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combined Strength-Endurance Circuit Training (Experimental)
  Interventions: Other: Strength-Endurance Training
- Endurance Circuit Training (Active Comparator)
  Interventions: Other: Endurance Training
- Control Group (No Intervention)

INTERVENTIONS:
Other: Strength-Endurance Training — The intervention for the experimental Strength-Endurance group includes warm-up, three laps of strength and endurance exercises and cool-down.
  The training program lasts 3 months and includes two 1-hour training sessions per week, for a total of 24 sessions.
  Arms: Combined Strength-Endurance Circuit Training
Other: Endurance Training — The intervention for the control Endurance training group includes warm-up, three laps of endurance exercises and cool-down. The training program lasts 3 months and includes two 1-hour training sessions per week, for a total of 24 sessions.
  Arms: Endurance Circuit Training

SUMMARY:
The goal of this clinical trial is to determine whether adding strength training to aerobic training has a comparable or greater effect on the clinical status of Parkinson's disease patients than a standalone aerobic training.

- Does combined strength-endurance circuit training provide added benefits to physical performance, disease severity, blood biomarkers, and quality of life in PD patients compared to standalone aerobic training?

Participants will:

* undergo outcome measurements before and after the 12-week intervention and a 3-month follow-up measurement,
* visit the clinic twice a week for 1-hour training sessions.
* selected patients will be given a smartwatch with a pedometer that will count their average number of steps before, during and after the training period

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* diagnosis of idiopathic Parkinson´s disease
* Hoehn-Yahr Scale ≤ 2,5
* stable dopaminergic medication

Exclusion Criteria:

* age ≥75 years
* Hoehn-Yahr Scale ≥ 2,5
* deep brain stimulation
* presence of freezing
* Camptocormia
* inability to walk without support
* inability to perform study procedures
* limiting co-morbidities
* attendance at training sessions below 70%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Movement Disorders Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II. and III. | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
  The maximum total UPDRS score is 272, indicating the worst possible disability from PD. The minimum total score is 0, indicating no disability from PD. Improvement greater than (-4.9) points or worsening more than (+4.2) points on MDS-UPDRS II+III represent a minimal clinically important difference.

SECONDARY OUTCOMES:
One Repetition Maximum (1RM) | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
  One Repetition Maximum in strength training is the maximum weight that can be lifted once while maintaining the correct lifting technique. It will be measured using a leg press machine for the lower extremities and a dumbbell chest press for the upper extremities.
Timed Up and Go Test (TUG) | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
  Mean TUG score for Non-falling PD patients on medication is 7.94 (2.15) seconds. MCID is 3.5 seconds.
Blood irisin levels | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
Cardiopulmonary Exercise Testing | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
The Parkinson's Disease Questionnaire (PDQ-39) | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
  The minimum score is 0, while the maximum score is 100. A higher score indicates a lower QoL.
Blood brain-derived neurotrophic factor levels | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
Blood cytokine levels | From enrollment to the end of treatment at 12 weeks and 12 weeks after the end of treatment (Follow-up)
Average number of steps | Average number of steps in the period before training (6 months), during the training period (3 months), period after training (3 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology and Centre of Clinical Neuroscience First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD), including the study protocol, statistical analysis plan, informed consent form, and clinical study report, will be made available upon reasonable request to qualified researchers, but will not be publicly accessible.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD will be shared with all qualified researchers upon reasonable request sent to a contact email.

REFERENCES:
- [Background] Corcos DM, Robichaud JA, David FJ, Leurgans SE, Vaillancourt DE, Poon C, Rafferty MR, Kohrt WM, Comella CL. A two-year randomized controlled trial of progressive resistance exercise for Parkinson's disease. Mov Disord. 2013 Aug;28(9):1230-40. doi: 10.1002/mds.25380. Epub 2013 Mar 27. PMID 23536417
- [Background] Kam TI, Park H, Chou SC, Van Vranken JG, Mittenbuhler MJ, Kim H, A M, Choi YR, Biswas D, Wang J, Shin Y, Loder A, Karuppagounder SS, Wrann CD, Dawson VL, Spiegelman BM, Dawson TM. Amelioration of pathologic alpha-synuclein-induced Parkinson's disease by irisin. Proc Natl Acad Sci U S A. 2022 Sep 6;119(36):e2204835119. doi: 10.1073/pnas.2204835119. Epub 2022 Aug 31. PMID 36044549
- [Background] Shi X, Gu Q, Fu C, Ma J, Li D, Zheng J, Chen S, She Z, Qi X, Li X, Wu S, Wang L. Relationship of irisin with disease severity and dopamine uptake in Parkinson's disease patients. Neuroimage Clin. 2024;41:103555. doi: 10.1016/j.nicl.2023.103555. Epub 2023 Dec 15. PMID 38134742
- [Background] Gamborg M, Hvid LG, Dalgas U, Langeskov-Christensen M. Parkinson's disease and intensive exercise therapy - An updated systematic review and meta-analysis. Acta Neurol Scand. 2022 May;145(5):504-528. doi: 10.1111/ane.13579. Epub 2022 Jan 8. PMID 34997759